CLINICAL TRIAL: NCT04485936
Title: Prospective, Single Center, Open-labeled Single Arm Study of Evaluation of the Effect of Tulip Device on Gastric Emptying Rate in Healthy Subjects
Brief Title: Evaluation of the Effect of Epitomee Device on Gastric Emptying Rate in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Epitomee medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRT-05-030
Record Dates: First submitted 2018-07-09; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epitomee Device (Experimental): the participants receive the device which is non-surgical, non-pharmacologic, medical Device designed to enhance the feeling of early satiation and prolonged satiety
  Interventions: Device: Epitomee Device

INTERVENTIONS:
Device: Epitomee Device — medical Device designed to enhance the feeling of early satiation and prolonged satiety

SUMMARY:
Evaluation of the effect of Epitomee Device on Gastric Emptying Rate in healthy subjects

DETAILED DESCRIPTION:
The participants will be enrolled in one investigational site. Subjects meeting eligibility criteria will undergo a gastric emptying test using gastric scintigraphy before any treatment (baseline).

Following the scintigraphy, the subjects will receive Tulip Device treatment - 2 capsules/day.

After repeated capsule intake for either 4 or 11 or 28 days, the subjects will undergo additional gastric emptying test with a capsule intake prior to the test meal.

ELIGIBILITY:
Inclusion Criteria:

1. 21 ≤ Age <65 years
2. 20 < BMI ≤ 40 kg/m2
3. Healthy subject
4. Subject is able and willing to give informed consent
5. Subject is able and willing to participate in the study and follow protocol procedures

Exclusion Criteria:

1. Significant swallowing disorders or difficulty swallowing
2. Suspected GI strictures, fistulas or other GI track obstructions
3. Crohn's disease or diverticulosis
4. Recent GI surgery
5. History of long-standing undigested food in the stomach
6. Known ulcer disease
7. Organic disease associated with gastroparesis such a Parkinson's disease, cerebrovascular accident, neuromuscular disease or eating disorder
8. Presence of a gastrostomy tube or gastric outlet obstruction
9. History or evidence of any active liver disease
10. Allergy to eggs
11. Treatment with anticholinergic or prokinetic agents
12. Treatment with proton-pump inhibitors
13. Hypothyroidism, hyperthyroidism or taking thyroid hormone deficiency drugs (such as L-thyroxine)
14. Prediabetes or Diabetes
15. Any history or evidence of significant cardiac, renal, neurologic, pulmonary, gastrointestinal, hematologic abnormality, chronic hepatic disease or any other disease or symptom which in the judgment of the investigator would interfere with the study or confound the results
16. Pregnancy or breastfeeding
17. Currently participating in an ongoing clinical study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of Epitomee device on Gastric half-emptying time | 10 days
  Change in Gastric half-emptying time

CONTACTS AND LOCATIONS:
Overall Officials: Haim Shirin, MD, Principal Investigator — The Kamila Gonczarowski Institute of Gastroenterology Assaf Harofeh Medical Center,
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participants data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within six months of study completion